CLINICAL TRIAL: NCT01823523
Title: Orthognathic Surgery and Postoperative Antibiotic Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Center for Oral and Maxillofacial Surgery (Other)
Responsible Party: Principal Investigator, Dr. Curtis Gregoire, Dr. Curtis Gregoire Oral and Maxillofacial Surgeon, Atlantic Center for Oral and Maxillofacial Surgery
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ACOMFS-Orthognathic
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Dentofacial Deformity
MeSH Terms: conditions — Dentofacial Deformities | interventions — Cefazolin; Cephalexin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefazolin, Cephalexin, Clindamycin (Active Comparator): Group will be receiving 1 day of IV cefazolin or clindamycin followed by 2 days of oral cephalexin or clindamycin
  Clindamycin will be used in patients with allergy
  Interventions: Drug: Cefazolin, Cephalexin, Clindamycin
- cefazolin, clindamycin, placebo (Placebo Comparator): Group will receive 1 day IV cefazolin, or clindamycin followed by 2 days of oral placebo
  clindamycin will be used if patient has allergy
  Interventions: Drug: Cefazolin, Cephalexin, Clindamycin

INTERVENTIONS:
Drug: Cefazolin, Cephalexin, Clindamycin
  Other Names: Ancef, Keflex, Dalacin C

SUMMARY:
Currently there is debate in the literature as to the recommended length of postoperative antibiotics in patients undergoing orthognathic surgery. The investigators plan to investigate using a randomized controlled trial the comparison between a 1 day and 3 day regimen of antibiotics and the effects on post operative infection.

DETAILED DESCRIPTION:
Capital Health Research Ethics Board Orthognathic Surgery and Postoperative Antibiotic Use Protocol

Background, Rationale and Statement of Research Question(s):

Surgical site infection is a potential problem with any surgical procedure. Surgical procedures done through the oral cavity are at a higher risk due to the presence of bacterial pathogens. Orthognathic surgery, involves incising through oral mucosa and creating osteotomies in underlying bony structures. Of the potential complications that can arise from this surgery, post operative infection (POI) is the most common. POI can have a significant impact on surgical outcomes and are associated with an increased cost to the health care system. The literature is quite clear on the benefits of presurgical prophylactic antibiotics in reducing the rate of post operative surgical site infections.1 Currently there is conflicting literature as to the recommended length patients should receive antibiotics during the postoperative course, and the majority of studies have small sample sizes.2,3

Orthognathic surgery is considered a clean-contaminated surgery with a suspected POI rate of 10-15%.2 In 1999 Bentley et. al conducted a randomized control trial comparing 1day vs 5day regimen of antibiotics following orthognathic surgery.4 This trial was stopped due to the drastic difference seen between the two groups, 6.7% in the 5 day course compared with 60% seen in the 1 day group.4 This data varies greatly from the rates of infection that the investigators have seen in their department using a 1 day course of antibiotics. Chow et al. in 2007 did a retrospective chart review of complications seen in orthognathic surgery. They found the rate of infection was significantly decreased by continuing antibiotics in the post operative course when compared to using only one prophylactic dose. They found the infection rates to be 17.3% with a single preoperative IV dose, 5.1% with a pre-operative dose and 2 days post-operative, and 7.7% with a pre-operative dose and 3 days of post-operative antibiotics.5 They also found no significant difference in rates of infection comparing 2 days and up to 14 days.5 A meta-analysis by Danda et al. in 2011 found that a regimen consisting of a single dose of preoperative antibiotics followed with an extended term postoperatively is the most effective in decreasing surgical site infections. They found the incidence decreased by 3.2 times, with the greatest effect noted with administration for 2 days.2 Even in this meta-analysis the average number of patients in each of the 8 studies was 67, with the total number of patients included being 532.2 This shows the need for randomized controlled studies with large sample sizes in order to determine the best antimicrobial regimen for these patients. The majority of studies investigating the rates of infection in orthognathic surgery use penicillin as the antibiotic of choice due to its spectrum of coverage for oral microbes and it is reasonably tolerated by patients.2,4-8 In the investigators department cefazolin is the antibiotic of choice and lower rates of infection have been observed compared to penicillin. The investigators suspect the lower rates of infection with cefazolin is due to the increased gram negative coverage and better resistance to beta lactamases. This has influenced the investigators decision to use first generation cephalosporins instead of penicillin as first line antimicrobials. In patients allergic to penicillin, clindamycin is used. The criteria for diagnosis of infection will follow the CDC guidelines for SSI. The primary outcome is to determine if there is any benefit to extending antimicrobials in the postoperative course following orthognathic surgery. Secondary outcomes include comparing the rates of infection between cefazolin/cephalexin groups and the clindamycin groups, and the rate of infection with different surgical procedures.

Currently at the CDHA the standard perioperative antimicrobial regimen for orthognathic surgery patients is one preoperative prophylactic dose of 2g of IV cefazolin followed by 1g IV every 8 hrs for 3 doses. Patients with an allergy to penicillin receive one preoperative prophylactic dose of IV Clindamycin 600mg, followed by 600mg IV every 8 hrs for 3 doses.

The investigators plan to conduct a double blind randomized controlled trial comparing the effect of a single day of post operative antibiotics with an extended 3 day course of antimicrobials on the infection rate. Both groups will receive an IV prophylactic dose followed by 3 IV doses postoperatively. Group 1 will then receive PO antibiotics for 2 subsequent days following IV treatment, and group 2 will receive a PO placebo.

A placebo will be used in order to blind the two groups so that the patient, surgeon and investigators are not aware of which patients are receiving the extended regimen of antibiotics. This will avoid potential bias in the patient report of symptoms or side effects, and the surgeon's bias in diagnosis of surgical site infection.

Subject Selection:

All patients over the age of 16 years undergoing orthognathic surgery at the QEII VG hospital are eligible to participate in the study. All surgeons operating at the VG site have been asked to include their patients in this study. These include patients undergoing either isolated Lefort I osteotomy, bilateral sagittal split osteotomies, functional genioplasties, or any combination of the three procedures. Wisdom teeth, if present, will also be extracted at the time of the surgery. Exclusion criteria include use of antibiotics in the past 2 weeks, active oral or odontogenic infection, significant medical condition, or if the patient is immunocompromised. All patients will have history and physical examination, CBC, INR/PTT, electrolytes as well as a radiographic evaluation prior to surgery. A power analysis was done to determine the required patient sample size for this study. This was done using a 5% change in infection as clinically significant and type I error of 0.05 with 0.90 power. The sample size required would be 397 patients. The investigators would like to enroll as many as possible over the next 2 years and anticipate to enroll approximately 500 patients. Study enrollment will finish in 2 years time from starting date, unless required sample size has not been met at which time it may be decided to extend length.

Research Plan:

All patients enrolled in the study will receive the standard preoperative IV prophylactic antibiotic, followed by 3 IV doses postoperatively. The patients will be randomly allocated to either the placebo or the antibiotic group at their presurgical assessment appointment. This allocation will be done by a clinical nurse, patients will be given a study patient number and handed a envelope from a folder that has been mixed sufficiently, inside this envelope will be a paper with an A or B denoting to the Shoppers Drug Mart pharmacy on the main floor of the VG hospital to dispense the according bottle they are to receive. This will be recorded beside their study number, and not be unblinded until the study is concluded. Blinding is important to avoid bias in assessment of infection by the surgeons, and to avoid bias in reporting of symptoms of either infection or side effects from the antibiotics. Following the completion of the IV antibiotic regimen, group 1 will receive oral cephalexin or clindamycin four times per day for 2 days and group 2 will receive a placebo four times per day for 2 days. All patients will also be sent home with specific oral hygiene instructions in addition to chlorhexidine 0.12% rinse to be used for 2 weeks postoperatively.

Patients will be assessed for signs of infection and recovery progress daily during hospital stay and during regular recall visits at 2 weeks and 4 weeks following discharge. There is no additional time requirements or cost to the patient by participating in this study. The diagnosis of infection will be made according to the CDC criteria of surgical site infection which include: purulent drainage, wound culture for known pathogen, at least one of signs or symptoms of infection (pain, tenderness, localized swelling, redness or heat)1.

The patient may withdrawl from the study at any time. A patient may be removed from the study if there is a significant change in the patients medical condition. An interm review of the rates of infection will be done and if the data demonstrates an increase risk to patients participating in study, the study will be stopped and unblinded.

All adverse events, serious adverse events, adverse drug reations will be reported to the Oral Maxillofacial Surgery Department and the patient will be assessed by the resident or attending surgeon.

Analysis of Data

All of the data will be organized and pooled according to each specific group. Following the study the blinding will be undone, and the primary outcome investigating the rate of infection will be analyzed in each of the four groups, 1 day cefazolin, 3 day cefazolin/cephalexin, 1 day clindamycin, 3 day clindamycin. Each of the 1 day groups will be compared and the 3 day groups in order to determine if the length of time on antibiotic has an effect on the rate of infection. Then the 1 day group and 3 day groups will be compared for the different type of antibiotic to see if the type of antibiotic has bearing on the length required. These comparisons will be done using a chi squared formula to look for statistical significance. This analysis will also be used to compare rates of infection between the type of surgical procedures done. Each of the groups will also be analyzed for possible confounding factors including time of surgery, age, sex, and oral hygiene status.

Confidentiality

All data will be kept secure by the research team by storing it in a locked office filing cabinet, or on a password protected file on the secured hospital network. Only the investigators, and research nurse will have access to this data. Following the study, the data will be kept in a locked cabinet for at least 25 years as required by law.

Harms

As all patients will receive the standard current protocol used at the investigators center, with the test group receiving an addition 2 days of antibiotics. The risks associated with participation in the study are those seen from prolonged antibiotic use. These include allergic reactions ranging from rash to anaphylaxis, toxic reactions to kidney, liver, gastrointestinal and secondary infections from candida or resistant pathogens. If anaphylaxis occurs normal protocol will be followed for treatment and monitoring. In the event of other adverse events from the antibiotic it will be stopped and any secondary infections will be treated appropriately. In the case of post operative infection this will be treated with a 10 day course of appropriate antibiotics.

Benefits

Overall the benefit of this study is to determine the ideal length of postoperative antibiotics in preventing post operative surgical site infections in patients undergoing orthognathic surgery. The group receiving an extended course of antibiotics potentially may have a lower rate of infection. Conversely, the placebo group may have the same rate of infection and avoid potential side effects of extended antibiotic treatment.

Disclosure of Any Financial Compensation

There will be no monetary compensation for participation in this study. Either the antibiotic or the placebo will be provided to the patient at no cost.

References

1. National Center for Infectious Diseases, Mangram AJ, Horan TC, Pearson ML, et. al. Guideline for Prevention of Surgical Site Infection, 1999. Infection Control and Hospital Epidemiology, 20:4:247- 278, 1999
2. Danda AK, Ravi P. Effectiveness of Postoperative Antibiotics in Orthognathic Surgery: A Meta-Analysis. J Oral Maxillofacial Surgery 69:2650-2656,2011
3. Tan SK, Lo J, Zwahlen RA. Perioperative Antibiotic Prophylaxis in Orthognathic Surgery: A Systematic Review and Meta-Analysis of Clinical Trials. Surg Oral Med Oral Pathology Oral Radiology Endodontics 112:19-27, 2011
4. Bentley KC, Head TW, Aiello GA. Antibiotic Prophylaxis in Orthognathic Surgery: A 1-Day Versus 5-Day Regimen. J Oral Maxillofacial Surgery 57:226-230.1999
5. Chow LK, Singh B, et al. Prevalence of Postoperative Complications After Orthognathic Surgery: A 15year Review. J Oral Maxillofacial Surgery 65:984-992, 2007
6. Ruggles JE, Hann JR, Antibiotic Prophylaxis in Intraoral Orthognathic Surgery. J Oral Maxillofacial Surgery 42:797-801, 1984.
7. Fridrich KL, Partnoy BE, Zeitler DL. Prospective analysis of Antibiotic Prophylaxis for Orthognathic Surgery. International Journal Adult Orthodontic and Orthognathic Surgery 9:129-131, 1994
8. Jansisyanont P, Sessirisombat S, Sastravaha P, Bamroong P, Antibiotic Prophylaxis for Orthognathic Surgery: A Prospective, Comparative, Randomized Study between Amoxicillin-Clavulanic Acid and Penicillin. J Med Association Thailand 11: 1726-31, 2008.

Advertisements

No advertisements will be used for enrollment in this study.

Additional Considerations

Funding has been provided by the Canadian Association of Oral and Maxillofacial Surgery.

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old undergoing orthognathic surgery

Exclusion Criteria:

* Use of antibiotics in last 2 weeks, active oral or odontogenic infection, significant medical condition, immunocompromised

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Rate of infection | 4 weeks following surgery
  Investigation of the incidence of post operative infection following surgery in each of the two groups

SECONDARY OUTCOMES:
Side effect from antibiotic use | 4 weeks
  investigation of the incidence of side effects from an extended antibiotic regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Danda AK, Ravi P. Effectiveness of postoperative antibiotics in orthognathic surgery: a meta-analysis. J Oral Maxillofac Surg. 2011 Oct;69(10):2650-6. doi: 10.1016/j.joms.2011.02.060. Epub 2011 May 6. PMID 21549486
- [Background] Tan SK, Lo J, Zwahlen RA. Perioperative antibiotic prophylaxis in orthognathic surgery: a systematic review and meta-analysis of clinical trials. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Jul;112(1):19-27. doi: 10.1016/j.tripleo.2010.07.015. Epub 2010 Dec 17. PMID 21168350
- [Background] Bentley KC, Head TW, Aiello GA. Antibiotic prophylaxis in orthognathic surgery: a 1-day versus 5-day regimen. J Oral Maxillofac Surg. 1999 Mar;57(3):226-30; discussion 230-2. doi: 10.1016/s0278-2391(99)90664-x. PMID 10077192
- [Background] Chow LK, Singh B, Chiu WK, Samman N. Prevalence of postoperative complications after orthognathic surgery: a 15-year review. J Oral Maxillofac Surg. 2007 May;65(5):984-92. doi: 10.1016/j.joms.2006.07.006. PMID 17448852
- [Background] Ruggles JE, Hann JR. Antibiotic prophylaxis in intraoral orthognathic surgery. J Oral Maxillofac Surg. 1984 Dec;42(12):797-801. doi: 10.1016/0278-2391(84)90348-3. PMID 6594473
- [Background] Fridrich KL, Partnoy BE, Zeitler DL. Prospective analysis of antibiotic prophylaxis for orthognathic surgery. Int J Adult Orthodon Orthognath Surg. 1994;9(2):129-31. PMID 7989814
- [Background] Jansisyanont P, Sessirisombat S, Sastravaha P, Bamroong P. Antibiotic prophylaxis for orthognathic surgery: a prospective, comparative, randomized study between amoxicillin-clavulanic acid and penicillin. J Med Assoc Thai. 2008 Nov;91(11):1726-31. PMID 19127796